CLINICAL TRIAL: NCT04865172
Title: ECOCAPTURE@HOME: Program for the Assessment of Behavioural Markers of Apathy Under Real-life Conditions Aimed At Patients with Neurodegenerative Dementias and Their Caregivers
Brief Title: ECOCAPTURE for the Assessment of Apathy Under Real-life Conditions
Acronym: @HOME
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C20-23; 2020-A03305-34 (Registry Identifier: ID RCB)
Record Dates: First submitted 2021-03-24; First posted 2021-04-29 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Frontotemporal Dementia, Behavioral Variant; Alzheimer Disease
MeSH Terms: conditions — Pick Disease of the Brain; Alzheimer Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patient-caregiver dyads, patients with behavioural variant frontotemporal dementia: 20 patient-caregiver dyads, patients with behavioural variant frontotemporal dementia
  Interventions: Other: Remote collection of passive and active data for 28 consecutive days
- Patient-caregiver dyads, patients with Alzheimer disease: 20 patient-caregiver dyads, patients with Alzheimer disease
  Interventions: Other: Remote collection of passive and active data for 28 consecutive days
- Healthy control dyads: 20 healthy control dyads
  Interventions: Other: Remote collection of passive and active data for 28 consecutive days

INTERVENTIONS:
Other: Remote collection of passive and active data for 28 consecutive days — Passive sensor data: collected continuously for 28 days, from a multi-sensor wearable bracelet worn by each member of the dyad; Active questionnaire data: collected once a week during the four weeks of monitoring (and at the end of the 28 days for patient-caregiver dyads), from questionnaires filled by one partner of the dyad (for patient-caregiver dyads, this will be the caregiver) using a smartphone application.

SUMMARY:
ECOCAPTURE@HOME is a study which is currently being developed with the objective to capture the behavioral signature of apathy in everyday life context through remote monitoring of participants' behavior for about one month. Participants will not only be patients with apathy but also their spouse caregiver. Behavioral markers of apathy will be extracted from a combination of: 1/ objective physiological data from sensors on a bracelet worn by participants; 2/ subjective data filled by the caregiver through an application. Thus investigators will collect a pool of metrics and show they can measure three assumed behavioral markers of apathy (daytime activity, quality of sleep and emotional arousal), which in turn allow to predict caregiver's perception of the dyad's psychological state. The final goal is to lay the foundations for the development of a clinical tool for the remote follow-up of patient-caregiver couples.

DETAILED DESCRIPTION:
Apathy, a common neuropsychiatric symptom associated with dementia, has a strong impact on both patients' and caregivers' quality of life. In spite of its debilitating consequences, apathy is still poorly understood and hard to define or measure objectively. The overall objective of the ECOCAPTURE programme is to define a precise behavioural signature of apathy, assessed by a multi-modal and ecological approach. This protocol called "ECOCAPTURE@HOME" aims to validate a novel method for the remote measurement of behavioural markers of apathy. The final purpose of such a protocol being to improve the diagnosis and long-term follow-up of apathy.

Investigators plan to recruit 60 couples aged between 40 and 85 years old and divided into three groups of dyads: one group of 20 patient-caregiver dyads in which patients suffer from the behavioral variant of Fronto-Temporal Dementia (bvFTD), one group of 20 patient-caregiver dyads in which patients suffer from Alzheimer Disease (AD) and one group of 20 healthy control couples. All recruited dyads will be followed in their everyday life for 28 consecutive days via a multi-sensor wearable bracelet (worn by both partners of the dyad) collecting passive behavioural data. Active behavioural data will also be collected using questionnaires available on a smartphone application (completed by caregiver in patient-caregiver dyads). Investigators will thus validate a measurement model for three theoretical behavioural markers of apathy (i.e., daytime activity, quality of sleep and emotional arousal) using a pool metrics extracted from passive behavioural data (acceleration, electrodermal activity and blood volume pulse) completed by active behavioural data (describing behaviour at meals, wake and bedtime). Moreover, investigators will investigate this measurement model on both a daily and a monthly scale and will attempt to show that the measured behavioural markers of apathy can predict caregiver's perception of the dyad's psychological state (collected through questionnaires) on these two time-scales.

This project carries great potential to improve both patients' care and caregivers' social support.

ELIGIBILITY:
Inclusion Criteria for patients:

1. Diagnosis of bvFTD according to Rascovsky's international criteria for the bvFTD group / diagnosis of AD according to Dubois's international criteria for the AD group;
2. No evidence of any other cerebral pathology;
3. A Mini-Mental State Evaluation (MMSE) score superior or equal to 10 (to minimise the effect of confounding factors related to very severe cognitive impairment);
4. Aged between 40 and 85;
5. No evidence of any psychiatric condition and a Montgomery-Åsberg Depression Rating Scale (MADRS) score inferior to 20 (to avoid confusion between depression and apathy);
6. No evidence of excessive consumption of psychotropic drugs - for instance benzodiazepines, sleeping pills, etc. (due to their tranquilising effect);
7. No major physical disability disrupting mobility;
8. No heart pacemaker (which would compromise heart rate measuring).

Inclusion Criteria for caregivers and partners of healthy control dyads:

1. Aged between 40 and 85;
2. No evidence of any psychiatric condition;
3. A MADRS score inferior to 20;
4. No evidence of excessive consumption of psychotropic drugs;
5. No major physical disability disrupting mobility;
6. No heart pacemaker.

Exclusion Criteria:

1. Persons in detention by judicial or administrative decision
2. Person who is subject to a legal protection order
3. Person submitted to an exclusion period due to the participation to another research

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 patient-caregiver dyads with patients suffering from behavioral variant front-temporal dementia, 20 patient-caregiver dyads with patients suffering from Alzheimer disease, 20 healthy control dyads
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Acceleration (in g) | 28 days
  In all the dyads included in the study for a remote follow-up, investigators will collect the acceleration signal recorded by a bracelet (Empatica E4) including a 3-axis accelerometer, continuously for 28 days. Data of acceleration will be collected in both partners of the dyad.
Electrodermal activity (in microsiemens) | 28 days
  In all the dyads included in the study for a remote follow-up, investigators will collect the electrodermal activity signal recorded by a bracelet (Empatica E4) including an EDA sensor, continuously for 28 days. Data of electrodermal activity will be collected in both partners of the dyad.
Blood volume pulse (or relative blood flow) | 28 days
  In all the dyads included in the study for a remote follow-up, investigators will collect the blood volume pulse recorded by a bracelet (Empatica E4) including a photoplethysmogram (PPG) sensor, continuously for 28 days. Data of blood volume pulse will be collected in both partners of the dyad. Heart rate (number of beats per minute) can be derived from the blood volume pulse.
Bedtime and getting up time (Week 1) | once during the first week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete bedtime (using a drop-menu with hours and minutes) and getting up time next day. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Bedtime and getting up time (Week 2) | once during the second week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete bedtime (using a drop-menu with hours and minutes) and getting up time next day. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Bedtime and getting up time (Week 3) | once during the third week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete bedtime (using a drop-menu with hours and minutes) and getting up time next day. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Bedtime and getting up time (Week 4) | once during the fourth week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete bedtime (using a drop-menu with hours and minutes) and getting up time next day. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Meal times (Week 1) | once during the first week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete meal times (start time and end time, using a drop-menu with hours and minutes), including breakfast time, lunch time and dinner time. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Meal times (Week 2) | once during the second week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete meal times (start time and end time, using a drop-menu with hours and minutes), including breakfast time, lunch time and dinner time. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Meal times (Week 3) | once during the third week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete meal times (start time and end time, using a drop-menu with hours and minutes), including breakfast time, lunch time and dinner time. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Meal times (Week 4) | once during the fourth week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete meal times (start time and end time, using a drop-menu with hours and minutes), including breakfast time, lunch time and dinner time. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Autonomy for going to bed and getting up (Week 1) | once during the first week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete two questions about autonomy to go to bed and to get up: "Your partner went to bed / got up:". The answers are provided using a Visual Analogue Scale with "entirely at your initiative" at one end and "entirely at their own initiative" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Autonomy for going to bed and getting up (Week 2) | once during the second week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete two questions about autonomy to go to bed and to get up: "Your partner went to bed / got up:". The answers are provided using a Visual Analogue Scale with "entirely at your initiative" at one end and "entirely at their own initiative" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Autonomy for going to bed and getting up (Week 3) | once during the third week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete two questions about autonomy to go to bed and to get up: "Your partner went to bed / got up:". The answers are provided using a Visual Analogue Scale with "entirely at your initiative" at one end and "entirely at their own initiative" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Autonomy for going to bed and getting up (Week 4) | once during the fourth week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete two questions about autonomy to go to bed and to get up: "Your partner went to bed / got up:". The answers are provided using a Visual Analogue Scale with "entirely at your initiative" at one end and "entirely at their own initiative" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Signs of tiredness (Week 1) | once during the first week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete two questions about signs of tiredness: "Did your partner show signs of tiredness before going to bed / after getting up?". The answers are provided using a Visual Analogue Scale with "Yes, numerous signs of tiredness" at one end and "No, no signs of tiredness" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Signs of tiredness (Week 2) | once during the second week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete two questions about signs of tiredness: "Did your partner show signs of tiredness before going to bed / after getting up?". The answers are provided using a Visual Analogue Scale with "Yes, numerous signs of tiredness" at one end and "No, no signs of tiredness" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Signs of tiredness (Week 3) | once during the third week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete two questions about signs of tiredness: "Did your partner show signs of tiredness before going to bed / after getting up?". The answers are provided using a Visual Analogue Scale with "Yes, numerous signs of tiredness" at one end and "No, no signs of tiredness" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Signs of tiredness (Week 4) | once during the fourth week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete two questions about signs of tiredness: "Did your partner show signs of tiredness before going to bed / after getting up?". The answers are provided using a Visual Analogue Scale with "Yes, numerous signs of tiredness" at one end and "No, no signs of tiredness" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Involvement in the activities related to meal (Week 1) | once during the first week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete three questions (one for each meal: breakfast, lunch and dinner) about the partner's involvement in the activities related to meal: "How did you perceive your partner's involvement in activities related to breakfast/lunch/dinner". The answers are provided using a Visual Analogue Scale with "No involvement at all" at one end and "Large amount of involvement" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Involvement in the activities related to meal (Week 2) | once during the second week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete three questions (one for each meal: breakfast, lunch and dinner) about the partner's involvement in the activities related to meal: "How did you perceive your partner's involvement in activities related to breakfast/lunch/dinner". The answers are provided using a Visual Analogue Scale with "No involvement at all" at one end and "Large amount of involvement" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Involvement in the activities related to meal (Week 3) | once during the third week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete three questions (one for each meal: breakfast, lunch and dinner) about the partner's involvement in the activities related to meal: "How did you perceive your partner's involvement in activities related to breakfast/lunch/dinner". The answers are provided using a Visual Analogue Scale with "No involvement at all" at one end and "Large amount of involvement" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Involvement in the activities related to meal (Week 4) | once during the fourth week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete three questions (one for each meal: breakfast, lunch and dinner) about the partner's involvement in the activities related to meal: "How did you perceive your partner's involvement in activities related to breakfast/lunch/dinner". The answers are provided using a Visual Analogue Scale with "No involvement at all" at one end and "Large amount of involvement" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Usefulness of involvement in the activities related to meal (Week 1) | once during the first week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete three questions (one for each meal: breakfast, lunch and dinner) about the usefulness of the partner's involvement in the activities related to meal: "How did you perceive the usefulness of your partner's involvement in activities related to breakfast/lunch/dinner". The answers are provided using a Visual Analogue Scale with "Completely useless" at one end and "Very useful" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Usefulness of involvement in the activities related to meal (Week 2) | once during the second week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete three questions (one for each meal: breakfast, lunch and dinner) about the usefulness of the partner's involvement in the activities related to meal: "How did you perceive the usefulness of your partner's involvement in activities related to breakfast/lunch/dinner". The answers are provided using a Visual Analogue Scale with "Completely useless" at one end and "Very useful" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Usefulness of involvement in the activities related to meal (Week 3) | once during the third week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete three questions (one for each meal: breakfast, lunch and dinner) about the usefulness of the partner's involvement in the activities related to meal: "How did you perceive the usefulness of your partner's involvement in activities related to breakfast/lunch/dinner". The answers are provided using a Visual Analogue Scale with "Completely useless" at one end and "Very useful" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Usefulness of involvement in the activities related to meal (Week 4) | once during the fourth week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete three questions (one for each meal: breakfast, lunch and dinner) about the usefulness of the partner's involvement in the activities related to meal: "How did you perceive the usefulness of your partner's involvement in activities related to breakfast/lunch/dinner". The answers are provided using a Visual Analogue Scale with "Completely useless" at one end and "Very useful" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Autonomy of the involvement in the activities related to meal (Week 1) | once during the first week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete three questions (one for each meal: breakfast, lunch and dinner) about the autonomy of the partner's involvement in the activities related to meal: "If your partner did help you in the activities involved at breakfast/lunch/dinner, were these:". The answers are provided using a Visual Analogue Scale with "Completely at your initiative" at one end and "Completely at their own initiative" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Autonomy of the involvement in the activities related to meal (Week 2) | once during the second week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete three questions (one for each meal: breakfast, lunch and dinner) about the autonomy of the partner's involvement in the activities related to meal: "If your partner did help you in the activities involved at breakfast/lunch/dinner, were these:". The answers are provided using a Visual Analogue Scale with "Completely at your initiative" at one end and "Completely at their own initiative" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Autonomy of the involvement in the activities related to meal (Week 3) | once during the third week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete three questions (one for each meal: breakfast, lunch and dinner) about the autonomy of the partner's involvement in the activities related to meal: "If your partner did help you in the activities involved at breakfast/lunch/dinner, were these:". The answers are provided using a Visual Analogue Scale with "Completely at your initiative" at one end and "Completely at their own initiative" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Autonomy of the involvement in the activities related to meal (Week 4) | once during the fourth week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete three questions (one for each meal: breakfast, lunch and dinner) about the autonomy of the partner's involvement in the activities related to meal: "If your partner did help you in the activities involved at breakfast/lunch/dinner, were these:". The answers are provided using a Visual Analogue Scale with "Completely at your initiative" at one end and "Completely at their own initiative" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Quantity of interactions during meals (Week 1) | once during the first week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete three questions (one for each meal: breakfast, lunch and dinner) about the quantity of interactions with the partner during meals: "How would you consider the interactions between you and your partner during breakfast/lunch/dinner?". The answers are provided using a Visual Analogue Scale with "None at all" at one end and "Very numerous" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Quantity of interactions during meals (Week 2) | once during the second week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete three questions (one for each meal: breakfast, lunch and dinner) about the quantity of interactions with the partner during meals: "How would you consider the interactions between you and your partner during breakfast/lunch/dinner?". The answers are provided using a Visual Analogue Scale with "None at all" at one end and "Very numerous" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Quantity of interactions during meals (Week 3) | once during the third week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete three questions (one for each meal: breakfast, lunch and dinner) about the quantity of interactions with the partner during meals: "How would you consider the interactions between you and your partner during breakfast/lunch/dinner?". The answers are provided using a Visual Analogue Scale with "None at all" at one end and "Very numerous" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Quantity of interactions during meals (Week 4) | once during the fourth week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete three questions (one for each meal: breakfast, lunch and dinner) about the quantity of interactions with the partner during meals: "How would you consider the interactions between you and your partner during breakfast/lunch/dinner?". The answers are provided using a Visual Analogue Scale with "None at all" at one end and "Very numerous" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Quality of interactions during meals (Week 1) | once during the first week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete three questions (one for each meal: breakfast, lunch and dinner) about the quality of interactions with the partner during meals: "Your partner's emotional reactions to your interactions seemed:". The answers are provided using a Visual Analogue Scale with "Entirely inappropriate" at one end and "Entirely appropriate" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Quality of interactions during meals (Week 2) | once during the second week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete three questions (one for each meal: breakfast, lunch and dinner) about the quality of interactions with the partner during meals: "Your partner's emotional reactions to your interactions seemed:". The answers are provided using a Visual Analogue Scale with "Entirely inappropriate" at one end and "Entirely appropriate" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Quality of interactions during meals (Week 3) | once during the third week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete three questions (one for each meal: breakfast, lunch and dinner) about the quality of interactions with the partner during meals: "Your partner's emotional reactions to your interactions seemed:". The answers are provided using a Visual Analogue Scale with "Entirely inappropriate" at one end and "Entirely appropriate" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.
Quality of interactions during meals (Week 4) | once during the fourth week of the follow-up
  In all the dyads included in the study for a remote follow-up, investigators will collect information on the behaviour of one of the dyad's partners (the patient in patient-caregiver dyads) through a questionnaire completed once a week by the other partner (caregiver in patient-caregiver dyads) using an application installed on their smartphone. In particular, the questionnaire will require to complete three questions (one for each meal: breakfast, lunch and dinner) about the quality of interactions with the partner during meals: "Your partner's emotional reactions to your interactions seemed:". The answers are provided using a Visual Analogue Scale with "Entirely inappropriate" at one end and "Entirely appropriate" at the other end. Each week, all questions of the questionnaire will have to be completed at the same time in the application.

SECONDARY OUTCOMES:
Patient's apathy perceived by caregiver (day scale) | once a week during the 4 weeks of the follow-up
  The secondary outcome measures will be collected through questionnaires completed by the caregiver (only in patient-caregiver dyads) using a smartphone application. For the measure of patient's apathy perceived by caregiver on a day scale (once a week), caregivers have to complete one question: "How did you perceive your partner's level of apathy (= lack of ability to initiate activities) during the day?" using a visual analogue scale from "Very low" to "Very high".
Patient's apathy perceived by caregiver (month scale) | at the end of the 28-day follow-up
  The secondary outcome measures will be collected through questionnaires completed by the caregiver (only in patient-caregiver dyads) using a smartphone application. For the measure of patient's apathy perceived by caregiver on the month scale (at the end of the 28 days of follow-up), investigators use a validated questionnaire: Starkstein Apathy Scale (SAS) in caregiver's version (Starkstein et al., 1992). SAS score varies between 0 and 42, higher score meaning higher apathy.
Caregiver's burden (day scale) | once a week during the 4 weeks of the follow-up
  The secondary outcome measures will be collected through questionnaires completed by the caregiver (only in patient-caregiver dyads) using a smartphone application. For the measure of caregiver's burden on a day scale (once a week), caregivers have to complete one question: "How did you perceive the level of burden related to your partner's care during the day?" using a visual analogue scale from "Very low" to "Very high".
Caregiver's burden (month scale) | at the end of the 28-day follow-up
  The secondary outcome measures will be collected through questionnaires completed by the caregiver (only in patient-caregiver dyads) using a smartphone application. For the measure of caregiver's burden on the month scale (at the end of the 28 days of follow-up), investigators use a validated questionnaire: Zarit Burden Interview (ZBI) (Hébert et al., 2010). ZBI score varies between 0 and 48, higher score meaning higher perceived burden.
Caregiver's health-related quality of life (day scale) | once a week during the 4 weeks of the follow-up
  The secondary outcome measures will be collected through questionnaires completed by the caregiver (only in patient-caregiver dyads) using a smartphone application. For the measure of caregiver's quality of life on a day scale (once a week), caregivers have to complete one question: "How did you perceive your overall health state (physical and psychological) during the day?" using a visual analogue scale from "Very bad health state" to "Very good health state".
Caregiver's health-related quality of life (month scale) | at the end of the 28-day follow-up
  The secondary outcome measures will be collected through questionnaires completed by the caregiver (only in patient-caregiver dyads) using a smartphone application. For the measure of caregiver's quality of life on the month scale (at the end of the 28 days of follow-up), investigators use a validated questionnaire: Short Form 36 (SF36) (Stewart, 2007). The SF-36 consists of eight scaled scores on a 0-100 scale. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Levy, MD, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- ICM, Hôpital Salpêtrière, Paris, France

REFERENCES:
- [Derived] Godefroy V, Levy R, Bouzigues A, Rametti-Lacroux A, Migliaccio R, Batrancourt B. ECOCAPTURE@HOME: Protocol for the Remote Assessment of Apathy and Its Everyday-Life Consequences. Int J Environ Res Public Health. 2021 Jul 23;18(15):7824. doi: 10.3390/ijerph18157824. PMID 34360133